CLINICAL TRIAL: NCT03057951
Title: A Phase III Randomised, Double-blind Trial to Evaluate Efficacy and Safety of Once Daily Empagliflozin 10 mg Compared to Placebo, in Patients With Chronic Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: EMPagliflozin outcomE tRial in Patients With chrOnic heaRt Failure With Preserved Ejection Fraction (EMPEROR-Preserved)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.110; 2016-002278-11 (EudraCT Number)
Record Dates: First submitted 2017-02-16; First posted 2017-02-20 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 10 mg Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — once daily
  Other Names: JARDIANCE, JARDIANZ, GIBTULIO
  Arms: 10 mg Empagliflozin
Drug: Placebo — once daily
  Arms: Placebo

SUMMARY:
This is a study in adults with chronic heart failure. People with chronic heart failure may need to be hospitalised for their condition. Some people with chronic heart failure may eventually die from their condition. The purpose of the study is to find out whether a medicine called empagliflozin lowers the chances of patients having to go to hospital for heart failure and whether it improves their survival. The study is open to patients with a type of chronic heart failure called chronic heart failure with preserved ejection fraction.

Participants stay in the study until researchers have enough information about how effective empagliflozin is. It is expected that participants who enter at the very beginning of the enrolment period may be in the study for over 3 years, while participants who enter near the end of the enrolment period may be in the study for less than 2 years. The participants are put into 2 groups. It is decided by chance who gets into which group. One group gets empagliflozin tablets every day and the other group gets placebo tablets every day. Placebo tablets look like empagliflozin tablets but contain no medicine.

Participants visit the doctors regularly. During these visits, the doctors collect information about the participant's health. The doctors want to know how many patients had to go to hospital because of heart failure or who died from cardiovascular disease.

ELIGIBILITY:
Inclusion criteria:

* Male or female patient, age >= 18 years at screening. For Japan only: Age >=20 years at screening
* Patients with chronic HF (Chronic Heart Failure) NYHA (New York Heart Association classification) class II-IV and preserved EF (Ejection Fraction)(LVEF (Left Ventricular Ejection Fraction) > 40 %) and elevated NT-proBNP (N-terminal of the prohormone brain natriuretic peptide) > 300 pg/ml for patients without AF, OR > 900 pg/ml for patients with AF, analysed at the Central laboratory at Visit 1
* Structural heart disease within 6 months prior to Visit 1, OR documented HHF (Hospitalisation for Heart Failure) within 12 months prior to Visit 1
* Stable dose of oral diuretics, if prescribed
* Signed and dated written ICF (informed consent form)
* Further inclusion criteria apply

Exclusion criteria:

* Myocardial infarction, coronary artery bypass graft surgery or other major cardiovascular surgery, stroke or TIA (Transient Ischaemic Attack) in past 90 days prior to Visit 1
* Heart transplant recipient or listed for heart transplant
* Acute decompensated HF (Heart Failure)
* Systolic blood pressure (SBP) >= 180 mmHg at Visit 2.
* Symptomatic hypotension and/or a SBP < 100 mmHg
* Indication of liver disease,
* Impaired renal function, defined as eGFR (Estimated Glomerular Filtration Rate) < 20 mL/min/1.73 m2 (CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration Equation))cr or requiring dialysis
* History of ketoacidosis
* Current use or prior use of a SGLT (Sodium-glucose co-transporter) -2 inhibitor or combined SGLT-1 and 2 inhibitor
* Currently enrolled in another investigational device or drug trial
* Known allergy or hypersensitivity to empagliflozin or other SGLT-2 inhibitors
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Further exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5988 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (616):
- United States (135):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Heart Center Research, LLC, Huntsville, Alabama
  - University of California San Francisco, Fresno, California
  - La Mesa Cardiac Center, La Mesa, California
  - Purushotham, Akther & Roshan Kotha, MD Inc., La Mesa, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Merced Vein and Vascular Center, Merced, California
  - Valley Clinical Trials, Inc., Northridge, California
  - University of California Irvine, Orange, California
  - Covigilant Research, LLC, Riverside, California
  - University of California San Francisco, San Francisco, California
  - University of California, Torrance, California
  - Orange County Research Center, Tustin, California
  - Blue Coast Cardiology, Vista, California
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Integrated Heart Care, Boca Raton, Florida
  - Southeast Clinical Research, LLC, Chiefland, Florida
  - Morton Plant Mease Health Care, Clearwater, Florida
  - Accel Research Sites, DeLand, Florida
  - Integrative Research Associates, Fort Lauderdale, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Elite Clinical Research, Miami, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Orlando Health Inc., Orlando, Florida
  - Peninsula Research, Inc., Ormond Beach, Florida
  - Clearwater Cardiovascular Consultants, Safety Harbor, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Advent Health Medical Group, Tampa, Florida
  - Grady Clinical Research Center, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Cardiovascular Group PC, Lawrenceville, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Atlanta Heart Specialists, LLC, Tucker, Georgia
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Mount Sinai Hospital, Chicago, Illinois
  - Advocate Health and Hospitals Corporation, Naperville, Illinois
  - Captain James A. Lovell Federal Health Care Center, North Chicago, Illinois
  - Rockford Cardiovascular Associates, Rockford, Illinois
  - Midwest Cardiovascular Research and Education Foundation, Elkhart, Indiana
  - St. Francis Medical Group-Indiana Heart Physicians, Inc, Indianapolis, Indiana
  - Reid Hospital, Richmond, Indiana
  - Beacon Medical Group Clinical Research, South Bend, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - Norton Heart Specialists, Louisville, Kentucky
  - Research Integrity, LLC, Owensboro, Kentucky
  - Grace Research, LLC, Bossier City, Louisiana
  - Clinical Trials of America, LLC, Monroe, Louisiana
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Maine Research Associates, Lewiston, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - MedStar Health Research Institute, Baltimore, Maryland
  - Metropolitan Cardiovascular Consultants, Beltsville, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - East Mountain Medical Associates, PC, Great Barrington, Massachusetts
  - Alpena General Hospital, Alpena, Michigan
  - McLaren Northern Michigan Hospital, Petoskey, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - Jackson Heart Clinic, P.A., Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - St. Louis Heart and Vascular, P.C., St Louis, Missouri
  - Deaconess Billings Clinic Research Center, Billings, Montana
  - Bozeman Health Clinical Research, Bozeman, Montana
  - Nebraska Heart Institute, Grand Island, Nebraska
  - CHI Health Midlands, Papillion, Nebraska
  - Healthcare Partners LLC, Las Vegas, Nevada
  - Palm Research Center, Las Vegas, Nevada
  - Advanced Heart Care, LLC, Bridgewater, New Jersey
  - Garden State Heart Care, PC, Manalapan, New Jersey
  - Capital Cardiology Associates, PC, Albany, New York
  - Trinity Medical WNY, PC, Cheektowaga, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Cardiovascular Consultants, New Hyde Park, New York
  - Mount Sinai - PRIME, New York, New York
  - Harlem Cardiology, New York, New York
  - Laurelton Heart Specialist, PC, Rosedale, New York
  - Saratoga Clinical Research, LLC, Saratoga Springs, New York
  - Northwell Health, Southampton, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - CHEAR Center LLC, The Bronx, New York
  - Cardiac Care and Vascular Medicine, PLLC, The Bronx, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Kernodle Clinic West, Burlington, North Carolina
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Clinical Trials of America, Inc, Lenoir, North Carolina
  - VA Northeast Ohio Healthcare System, Cleveland, Ohio
  - Rama Research LLC, Marion, Ohio
  - South Oklahoma Heart Research Group, Oklahoma City, Oklahoma
  - Doylestown Health Cardiology, Doylestown, Pennsylvania
  - Lycoming Internal Medicine, Inc, Jersey Shore, Pennsylvania
  - Richard M Kastelic and Associates, Johnstown, Pennsylvania
  - York Hospital, WellSpan Health, York, Pennsylvania
  - Lowcountry Center for Veterans Research, Charleston, South Carolina
  - Palmetto Health, Columbia, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Palmetto Research Center, LLC, Spartanburg, South Carolina
  - Sanford Research, Sioux Falls, South Dakota
  - The Stern Cardiovascular Center, Germantown, Tennessee
  - Apex Cardiology/ Research Associates of Jackson, Jackson, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - Seton Heart Institute, Austin, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Soltero Cardiovascular Research Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of North Texas Health Science Center, Fort Worth, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Angiocardiac Care of Texas, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Biopharma Informatic, Inc. Research Center, Houston, Texas
  - Private Practice Leadership, LLC, Katy, Texas
  - Baylor Scott and White Health, Plano, Texas
  - Alpine Research Organization, Farmington, Utah
  - Cardiac Health Management Network, P.C., Chester, Virginia
  - Cardiology Consultants of Danville, Inc, Danville, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Medical College of Virginia Hospitals, Richmond, Virginia
  - Roanoke Heart Institute PLC, Roanoke, Virginia
  - Salem VA Medical Center, Salem, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Cardiology Associates of Bellin Health, Green Bay, Wisconsin
  - Meriter Wisconsin Heart, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aspirus Research Institute, Wausau, Wisconsin
- Argentina (39):
  - Hospital Interzonal General de Agudos Dr Jose Penna, Bahía Blanca
  - Hospital Italiano Regional del Sur, Bahia Blanca, Bahía Blanca
  - CIPREC, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Instituto Cardiovascular de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Glenny Corp. S.A. Bioclinica Argentina, Ciudad Autonoma Buenos Aires
  - Centro Médico Viamonte, Ciudad Autonoma de Bs As
  - Consultorios Asociados de Endocrinología e Invest Clínica, Ciudad Autonoma de BuenosAires
  - Sanatorio Güemes, Ciudad Autónoma de Bs As
  - Instituto Medico Elsa Perez SRL (IMEP), Ciudadela
  - Clinica Coronel Suarez SA, Coronel Suárez
  - Instituto de Cardiología de Corrientes, Corrientes
  - Sanatorio Mayo Privado SA, Córdoba
  - Centro de Investigaciones Clinicas Instituto del Corazon, Córdoba
  - Sanatorio Allende S.A., Córdoba
  - Clinica Privada Colombo- Fundacion Clinica Colombo, Córdoba
  - Instituto Médico DAMIC S.R.L., Córdoba
  - Hospital Privado, Córdoba
  - Hospital Italiano de La Plata, La Plata
  - Centro de Investigaciones Médicas, Mar del Plata
  - Hospital Privado de Comunidad, Mar del Plata
  - CER Instituto Médico, Quilmes
  - Instituto de Investigaciones Clínicas de Quilmes, Quilmes
  - Instituto de Investigaciones Clinicas de Rosario, Rosario
  - Instituto Medico Fundación Grupo Colaborativo Rosario, Rosario
  - Sanatorio Británico, Rosario
  - Sanatorio Plaza, Rosario
  - Instituto CAICI, Rosario
  - CORDIS S.A., Salta, Salta
  - Centro Cardiovascular Salta, Salta
  - Corporacion Medica de Gral. San Martin S.A., San Martín
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán
  - Instituto de Cardiología, San Miguel de Tucumán
  - Clinica Mayo, San Miguel de Tucumán
  - Centro Medico Luquez, San Vicente
  - Centro de Investigaciones Clínicas del Litoral, Santa Fe
  - Hospital "Dr. José Maria Cullen", Santa Fé
  - Clínica Olivos, Vicente López
  - CEMEDIC - Centro de Especialidades Medicas, Villa Luro
- Australia (13):
  - Pendlebury Research, Kotara, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - CORE Research Group, Milton, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Adelaide Medical Research, Ashford, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Heart and Vascular Research, Fullarton, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - The Northern Hospital, Epping, Victoria
  - Peninsula Private Hospital, Frankston, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - Mount Hospital, Perth, Western Australia
- Belgium (9):
  - C.H.U. de Charleroi, Charleroi
  - AZ Sint-Blasius, Dendermonde
  - Ziekenhuis Oost-Limburg - Campus Sint-Jan, Genk
  - AZ Maria Middelares, Ghent
  - Grand Hôpital de Charleroi, Gilly
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - La Louvière - UNIV CHU Tivoli, La Louvière
  - UZ Leuven, Leuven
  - Liège - HOSP CHR de la Citadelle, Liège
- Brazil (37):
  - FGM - Clínica Paulista de Doenças Cardiovasculares, Bela Vista
  - Hospital Felicio Rocho, Belo Horizonte
  - Hospital Vera Cruz, Belo Horizonte
  - L2IP -Instituto de Pesquisas Clínicas Ltda., Brasília
  - ICDF - Instituto de Cardiologia do Distrito Federal, Brasília
  - CECAP - Centro de Cardiologia Clínica, Brasília
  - Irmandade da Santa Casa de Misericordia de Curitiba, Campina Grande do Sul
  - Centro Especializado em Cardiol Loema Instituto de Pesq Clin, Campinas
  - IPECC - Instituto de Pesquisa Clínica de Campinas, Campinas
  - CAEP - Centro Avançado de Estudos e Pesquisas Ltda.,Campinas, Campinas
  - Hospital Universitário, Canoas
  - IPCEM - Instituto de Pesquisa Clínica para Estudos Multicêntricos - Universidade de Caxias do Sul, Caxias do Sul
  - Irmandade da Santa Casa de Misericórdia de Curitiba, Curitiba
  - Via Medica, Goiânia
  - HC-UFG - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia
  - ICM - Instituto do Coracao de Marilia, Marília
  - Hospital São Vicente de Paulo, Passo Fundo
  - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Centro de Pesquisas em Diabetes, Porto Alegre
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Instituto de Cardiologia Rio Grande do Sul, Porto Alegre
  - Hospital Agamenon Magalhaes, Recife
  - H.C.da Fac. de Medicina de Ribeirao Preto, Ribeirão Preto
  - Hospital Universitário Pedro Ernesto UERJ, Rio de Janeiro
  - CCBR - Rio de Janeiro - BR, Rio de Janeiro
  - Cardresearch Cardiologia Assistencial e de Pesquisas Ltda, Santa Efigênia
  - Pesquisare, Santo André
  - Praxis Pesquisa Médica, Santo André
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Hospital de Base - Fac Med de Sao Jose do Rio Preto, São José do Rio Preto
  - Centro de Pesquisa Clinica - CPCLIN, São Paulo
  - CDEC BRASIL - Centro de Desenvolvimento em Estudos Clínicos Brasil, São Paulo
  - CEPIC - Centro Paulista de Investigacao Clinica, São Paulo
  - Dr. Consulta, São Paulo
  - INCOR e Hospital das Clínicas da Universidade de São Paulo, São Paulo
  - CEDOES - Diagnóstico e Pesquisa,Vitória, Vitória
  - Santa Casa de Votuporanga, Votuporanga
- Canada (34):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Medical Arts Health Research Group, North Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - G.A. Research Associates Ltd, Moncton, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Brampton Cardio Pulmonary Clinic, Brampton, Ontario
  - Brampton Research Associates, Brampton, Ontario
  - JBN Medical Diagnostic Services Inc., Burlington, Ontario
  - Cambridge Cardiac Care Inc., Cambridge, Ontario
  - Dr. Saul Vizel, Cambridge, Ontario
  - Cardiovascular Contract Research Organization LTD, Greater Sudbury, Ontario
  - Curnew Medicine Professional Corporation, Hamilton, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - University Hospital (LHSC), London, Ontario
  - PACE (Partners in Advanced Cardiac Evaluation), Newmarket, Ontario
  - M Heffernan Medicine Professional Corp., Oakville, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Heart Health Institute, Scarborough Village, Ontario
  - Scarborough Cardiology Research, Scarborough Village, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - North York Diagnostic and Cardiac Centre, Toronto, Ontario
  - Mohan Babapulle Medicine Professional Medicine, Waterloo, Ontario
  - Dr. Louis C.H. Yao, York, Ontario
  - ViaCar Recherche Clinique Inc, Brossard, Quebec
  - ViaCar Recherche Clinique Inc, Greenfield Park, Quebec
  - Centre de Dépistage et Recherche Cardiovasculaire Rive-Sud, Longeuil, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Clinique Santé Cardio MC, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - IUCPQ (Laval University), Québec
- China (27):
  - Cardiovascular Institute and Fu Wai Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - First Hospital of Jilin University, Changchun
  - Hunan Provincial People's Hospital, Changsha
  - 2nd Xiangya Hospital of Central South University, Changsha
  - The Third Hospital of Changsha, Changsha
  - Dongguan People's Hospital, Dongguan
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - The First Afiliated Hospital, Sun Yet-sen University, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Haikou People's Hospital, Haikou
  - HaiNan Provincial People's Hospital, Haikou
  - The First Affiliated Hospital of Lanzhou University, Lanzhou
  - The Second Affiliated Hospital of Lanzhou Medical University, Lanzhou
  - The Affiliated Hospital of Southwest Medical University, Luzhou
  - Nanchang University Affiliated 3rd Hospital, Nanchang
  - First Hospital Affiliated with Nanjing Medical University, Nanjing
  - Huashan Hospital, Fudan University, Shanghai
  - General Hospital of Shenyang Military Region, Shenyang
  - Shengjing Hospital of China Medical University, Shenyang
  - Tianjin Union Medical Center Nankai University Affiliated Hospital, Tianjin
  - Tongji Hospital, Tongji University, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - First Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - Yanbian University Hospital, Yanji
  - the first people hospital of Yue Yang, Yueyang
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- Colombia (13):
  - Corazon IPS S.A.S., Barranquilla
  - Centro de Reumatologia y Ortopedia SAS, Barranquilla, Barranquilla
  - IPS Centro Cientifico Asistencia, Barranquilla
  - CardioColombia S.A.S., Bogota D.C
  - Endocare Research Institute, Bogotá
  - IPS Centro Medico Julián Coronel S.A., Cali
  - Fundación Valle del Lili, Cali
  - Centro de Investigaciones Clinicas S.A.S, Cali
  - Centro de Diagnostico Cardilogico, Cartagena
  - Centro cardiovascular Aristides, Cartagena
  - Fundación Cardiovascular de Colombia, Floridablanca
  - Asociacion IPS Medicos Internistas de Caldas, Manizales
  - Promotora Medica Las Americas SA, Medellín
- Czechia (30):
  - Poliklinika Humanitas, Bílovec
  - Internal and Cardiology Practice, MUDr. Karel Kamenik, Brno, Brno
  - MUDr. Alexandra Ludkova, Brno
  - University Hospital Brno, Brno
  - Vojenska nemocnice Brno, Brno
  - Nemocnice Milosrdnych bratri, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Univ.Hosp U Svate Anny, I.Internal Clinic-Cardiology,Brno, Brno
  - Edumed s.r.o, Broumov
  - MUDr. Jan Hubac, s.r.o. Kardiologicka ambulance, Chrudim
  - Hospital Frydek Mistek, Frýdek-Místek
  - Nemocnice Havlickuv Brod p.o., Havlíčkův Brod
  - Gepamed s.r.o., Pulm. Outpat. Office, Hradec Kralove, Hradec Králové
  - KardioLouny s.r.o., Louny
  - InterKardioML s.r.o., Mariánské Lázně
  - Zdenek Vomacka, Olomouc
  - PV-Kardiologie s.r.o., Pardubice
  - Vseobecna fakultni nemocnice V Praze, Prague
  - Institute for Clinical and Experimental Medicine, Prague
  - University Hospital Motol, Prague
  - Corintez s.r.o., Prague
  - University Thomayer's Hospital, Praha 4 - Krc
  - Kardio Vaclavik s.r.o., Přerov
  - Kardiologicka ambulance MUDr. Ferkl s.r.o., Trutnov
  - Nemocnice Trebic p.o., Třebíč
  - Kardiologicka ambulance, Třemošná
  - Clinical Trials Services s.r.o, Uherské Hradiště
  - Cardiology Private Practice, Uničov
  - Angiocor s.r.o, Zlín
  - KIGE s.r.o, Znojmo
- Germany (33):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Praxis Dr. Rieker, Berlin, Berlin
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinikum Bielefeld gGmbH, Bielefeld
  - Augusta-Kranken-Anstalt gGmbH, Bochum
  - Praxis Dr. Menzel, Dessau
  - St. Johannes Hospital Dortmund, Dortmund
  - Städtisches Klinikum Dresden, Dresden
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Studienzentrum Bocholderstraße, Essen
  - ClinPhenomics GmbH & Co KG, Frankfurt, Frankfurt
  - Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Asklepios Klinik Langen-Seligenstadt GmbH, Langen
  - Märkische Gesundheitsholding GmbH & Co. KG, Klinikum Lüdenscheid, Lüdenscheid
  - Praxis Dr. Sarnighausen, Lüneburg, Lüneburg
  - Katholisches Klinikum Mainz, Mainz
  - Gemeinschaftspraxis Drs. Kohler/Salbach, Mannheim, Mannheim
  - Deutsches Herzzentrum München, München
  - Gemeinschaftspraxis Dres Haggenmiller/Jeserich, Nuremberg
  - Kardiologische Praxis Papenburg, Papenburg
  - Universitätsklinikum Regensburg, Regensburg
  - Praxis Dr. Stenzel, Riesa, Riesa
  - Zentrum für Klinische Forschung, Wangen
  - Josephs-Hospital Warendorf, Warendorf
  - Kardiologische Praxis, Wermsdorf, Wermsdorf
  - Petrus-Krankenhaus, Wuppertal
- Hungary (20):
  - Lausmed Kft. Outpatient Unit of Internal Medicine, Baja
  - Belgyogyaszati es Kardiologiai Maganrendelo, Békéscsaba
  - Budai Irgalmasrendi Korhaz, Budapest
  - Clinexpert Kft., Budapest
  - Bajcsy-Zsilinszky Hospital and Clinic, Budapest
  - Semmelweis University, Budapest
  - Milit.Hosp.-State Health Cent., Budapest
  - Uzsoki Street Hospital, Budapest, Budapest
  - Nehezlegzes Ambulancia, Debrecen
  - University Debrecen Hospital, Debrecen
  - Bugat Pal Hospital, Gyongyos, Gyöngyös
  - Studium Egeszseghaz Kft., Kalocsa
  - Selye Janos Hospital Komarom, Komárom
  - Dorottya Kanizsai Hospital, Nagykanizsa
  - Medifarma-98 Kft., Nyíregyháza
  - Dr. Nagy Laszlo Kardiologiai Maganrendeles, Orosháza
  - University of Pecs, Pécs
  - Da Vinci Private Clinic, Pécs
  - Fejer County Saint George University Teaching Hospital, Székesfehérvár
  - Veszpremi Sziv es Egeszseg Centrum, Veszprém
- India (15):
  - Doctor Jivraj Mehta Smarak Health Foundation, Ahmedabad
  - Kamalnayan Bajaj Hospital, Aurangabad
  - Narayana Institute of Cardiac Sciences, Bangalore
  - Rajarajeswari Medical College, Bengaluru
  - Madras Medical Mission,, Chennai
  - Apollo Speciality Hospital, Chennai
  - GNRC Hospital, Guwahati
  - Medanta-The Medicity, Gūrgaon
  - B.M. Birla Heart research Centre, Kolkata
  - Vijan Cardiac and Critical Care Centre, Nashik
  - Siddhi Hospital, Nashik
  - GB Pant Hospital, New Delhi
  - Fortis Escorts Heart Institute, New Delhi
  - Sir Gangaram Hospital, New Delhi
  - Batra Hospital and Medical Research Centre, New Delhi
- Italy (13):
  - Azienda Ospedaliera G. Rummo, Benevento
  - ASST Papa Giovanni XXIII - A.O. Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna, Cona (FE)
  - Ospedale della Val di Chiana Santa Margherita, Cortona
  - Milano Fondazione IRCCS Ca'Granda-Ospedale Maggiore Policlinico, Milan
  - Centro Cardiologico Monzino-IRCCS, Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - AOU Policlinico Umberto I, Roma
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
  - Istituto Clinico Humanitas, Rozzano (MI)
  - IRCCS Gruppo Multimedica, Sesto San Giovanni (MI)
  - Azienda Servizi Sanitari 1 Triestina, Trieste
- Japan (65):
  - Kasugai Municipal Hospital, Aichi, Kasugai
  - Japanese Red Cross Nagoya Daini Hospital, Aichi, Nagoya
  - Chiba Heart Clinic, Chiba, Chiba
  - Kimitsu Chuo Hospital, Chiba, Kisarazu
  - Seikeikai New Tokyo Heart Clinic, Chiba, Matsudo
  - Ehime Prefectural Central Hospital, Ehime, Matsuyama
  - Matsuyama Shimin Hospital, Ehime, Matsuyama
  - Uwajima City Hospital, Ehime, Uwajima
  - Fukuiken Saiseikai Hospital, Fukui, Fukui
  - Fukuoka University Chikushi Hospital, Fukuoka, Chikushino
  - Fukuokaken Saiseikai Futsukaichi Hospital, Fukuoka, Chikushino
  - Saiseikai Fukuoka General Hospital, Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Steel Memorial Yawata Hospital, Fukuoka, Kitakyushu
  - Japan Community Health Care Organization Kyushu Hospital, Fukuoka, Kitakyushu
  - Shirakawa Kosei General Hospital, Fukushima, Shirakawa
  - Ogaki Municipal Hospital, Gifu, Ogaki
  - Chuno Kosei Hospital, Gifu, Seki
  - Fukuyama City Hospital, Hiroshima, Fukuyama
  - Shobara Red Cross Hospital, Hiroshima, Shobara
  - Matsuda Cardiovascular Clinic, Hokkaido, Sapporo
  - Teine Keijinkai Clinic, Hokkaido, Sapporo
  - Tomakomai City Hospital, Hokkaido, Tomakomai
  - Otaru Kyokai Hospital, Hokkaido,Otaru
  - Hyogo Prefectural Amagasaki General Medical Center, Hyogo, Amagasaki
  - Hyogo Brain and Heart Center, Hyogo, Himeji
  - National Hospital Organization Kobe Medical Center, Hyogo, Kobe
  - Mito Medical Center, Ibaraki, Higashiibaraki-gun
  - Tokushukai Koga General Hospital, Ibaraki, Koga
  - National Hospital Organization Kanazawa Medical Center, Ishikawa, Kanazawa
  - Mitoyo General Hospital, Kagawa, Kanonji
  - Kagawa Prefectural Central Hospital, Kagawa, Takamatsu
  - Sekishinkai Second Kawasaki Saiwai Clinic, Kanagawa, Kawasaki
  - Yamamoto Clinic, Kanagawa, Sagamihara
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - Seiwakai Suizenji Touya Hospital, Kumamoto, Kumamoto
  - Kumamoto Rosai Hospital, Kumamoto, Yatsushiro
  - Omi Medical Center, Kusatsu
  - Uji-Tokushukai Medical Center, Kyoto, Uji
  - Sendai Kousei Hospital, Miyagi, Sendai
  - Sendai Tokushukai Hospital, Miyagi, Sendai
  - National Hospital Organization Sendai Medical Center, Miyagi, Sendai
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Hokushin General Hospital, Nagano, Nakano
  - Nagasaki Medical Center, Nagasaki, Omura
  - Oita Medical Center, Oita, Oita
  - Okayama City General Medical Center, Okayama, Okayama
  - Naha City Hospital, Okinawa, Naha
  - Nanbu Tokushukai Hospital, Okinawa, Shimajiri-gun
  - Urasoe General Hospital, Okinawa, Urasoe
  - Higashiosaka City Medical Center, Osaka, Higashiosaka
  - Kitano Hospital, Osaka, Osaka
  - Yodogawa Christian Hospital, Osaka, Osaka
  - Hokusetsu General Hospital, Osaka, Takatsuki
  - San-Ai Hospital, Saitama, Saitama
  - Kosekai Iwatsuki-minami Hospital, Saitama, Saitama
  - Tokushima Prefectural Central Hospital, Tokushima, Tokushima
  - National Hospital Organization Tokyo Medical Center, Tokyo, Meguro-ku
  - Ome Municipal General Hospital, Tokyo, Ome
  - Tokyo Rosai Hospital, Tokyo, Ota-ku
  - Sekino Hospital, Tokyo, Toshima-ku
  - Minami Wakayama Medical Center, Wakayama, Tanabe
  - Kanmon Medical Center, Yamaguchi, Shimonoseki
- Mexico (14):
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Centro de Investigacion Biomedica y Farmaceutica, S.C., Distrito Federal
  - Hospital Ramon Garibay, Guadalajara
  - Diseño y Planeación en Investigación Médica SC, Guadalajara
  - Unidad de Investigacion Clinica Cardiometabolica de Occident, Guadalajara
  - Cardiologia Clinica e Intervencionista, Guadalajara
  - Centro de Investigación Clinica Acelerada, S.C., México
  - CEDOPEC-Ctro Esp en Diab, Obesidad y Prev de Enf Cardiovasc, México
  - Instituto Cardiovascular de Monclova, S de RL de CV, Monclova
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Nuevo León
  - Centro Integral Medico SJR S.C., San Juan del Río
  - Cardioarritmias e Investigación S.C, San Luis Potosí City
  - Centro de Investigacion Cardiovascular y Metabolica, Tijuana
  - Centro de Investigacion Medica Alberto Bazzoni S.A. de C.V., Torreón
- Netherlands (20):
  - Ziekenhuisgroep Twente locatie Almelo, Almelo
  - BovenIJ Ziekenhuis, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Locatie West, Amsterdam
  - Amsterdam UMC Locatie VUMC, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Amsterdam UMC, Locatie AMC, Amsterdam
  - Rode Kruis Ziekenhuis Beverwijk, Beverwijk
  - Tergooiziekenhuizen locatie Blaricum, Blaricum
  - Amphia Ziekenhuis, Breda
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Universitair Medisch Centrum Groningen, Groningen
  - Zuyderland Medisch Centrum, Heerlen
  - Maastricht University, Maastricht
  - Diaconessenhuis Meppel, Meppel
  - St. Antonius ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Franciscus Gasthuis, Rotterdam
  - De Heel - Zaans Medisch Centrum, Zaandam
  - Gelre Ziekenhuis Zutphen, Zutphen
- Poland (35):
  - Univ. Clinic Hosp, Bialystok, Bialystok
  - KLIMED Marek Klimkiewicz, Bialystok
  - ClinicMed Badurski i wspolnicy Spolka Jawna, Bialystok, Bialystok
  - American Heart of Poland Sp. z o.o., Bielsko-Biala
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Polsko-Amerykanskie Kliniki Serca, Chorzów
  - American Heart of Poland Sp. z o.o., Dąbrowa Górnicza
  - Poradnia Kardiologiczna Jaroslaw Jurowiecki, Gdansk
  - University Clinical Center, Gdansk, Gdansk
  - Indywidualna Specjalistyczna Praktyka Lekarska, Gdynia
  - NZOZ Pro-Cordis Sopockie Centrum Bad. Kardiolog., Gdynia
  - Szpital Zakonu Bonifratow Sp. z o.o., Katowice
  - Specialistic Cardiology&Hypertension Out-patient Clin,Kielce, Kielce
  - Leszek Bryniarski Specialized Medical Cabinet, Krakow
  - Krakow Specialistic Hospital of John Paul II, Krakow
  - ETG Lodz, Lodz
  - Nzoz Salus, Lodz
  - Individual Specialized Practice, Lodz
  - Lowickie Cardiology Center, Lowicz
  - American Heart of Poland Sp. z o.o., Nysa
  - Medicome Sp. z o.o., Oświęcim
  - NZOZ HEUREKA, Piaseczno, Piaseczno
  - Specialized Practice Dr. Janusz Spyra, Ruda Śląska
  - Centrum Medyczne Medyk, Rzeszów
  - Lukmed Lukasz Wozniak, Siedlce
  - ETG Skierniewice, Skierniewice
  - KO-MED Centra Kliniczne Staszow, Staszów
  - The Provincial Polyclinical Hospital in Torun, Torun
  - American Heart of Poland Sp. z o.o., Tychy
  - American Heart of Poland Sp. z o.o., Ustroń
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
  - ETG Warszawa, Warsaw
  - 4. Military Clinical Hospital with Polyclinic SP ZOZ, Wroclaw
  - Zgierskie Center of Cardiology MED-PRO, Zgierz
  - Specialist Hospital J. Dietla NZOZ Specialized Clinic "Gemini", Żychlin
- Romania (13):
  - Spitalul Clinic De Urgenta "Prof. Dr. Agrippa Ionescu", Baloteşti
  - C.M.D.T.A. NEOMED, Brasov, Brasov
  - CMDTA Washington, Bucharest, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Emergency Clinical Hospital 'Sf. Panteliomon', Bucharest
  - Emergency University Hospital, Bucharest, Bucharest
  - Prof.C.C.Iliescu Hospital, National Institute of Cardiology, Bucharest
  - Spitalul Clinic "Prof. Dr. Theodor Burghele", Bucharest
  - Clinica Medicala Data Plus SRL, Bucharest
  - S.C Cardiomed S.R.L, Craiova
  - Spital Judetean Deva, Deva
  - S.C Medicali's S.R.L, Timișoara
  - Spitalul Clinic Judetean de Urgenta, Timisoara, Timișoara
- Singapore (4):
  - National University Hospital, Singapore
  - National Heart Center, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore
- South Africa (13):
  - Cardiology Clinical Research, Alberton
  - Iatros International, Bloemfontein
  - Universitas Hospital Cardiology Research, Bloemfontein
  - Corbod Research, Cape Town
  - TREAD Research, Cape Town
  - Tiervlei Trial Centre, Cape Town
  - Excellentis Clinical Trials, George
  - Clinresco, Johannesburg
  - Chris Hani Baragwanath Hospital: Cardiology Department, Johannesburg
  - MERC Research, Kempton Park
  - Into Research, Pretoria
  - Dr JM Engelbrecht, Somerset West
  - Clinical Projects Research, Worcester
- South Korea (13):
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Wonju Severance Christian Hosp, Wŏnju
- Spain (13):
  - Hospital Quiron. I.C.U., Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Sanitas CIMA, Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital La Paz, Madrid
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Virgen Macarena, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
- United Kingdom (8):
  - Barnet General Hospital, Barnet
  - University Hospital of Wales, Cardiff
  - Park & St Francis Surgery, Eastleigh
  - Wycombe General Hospital, High Wycombe
  - Glenfield Hospital, Leicester
  - St Bartholomew's Hospital, London
  - St Mary's Hospital, Newport
  - Morriston Hospital, Swansea

REFERENCES:
- [Derived] Ferreira JP, Packer M, Butler J, Vasques-Novoa F, Marques P, Pocock S, Filippatos G, Zannad F, Anker SD. Serum Magnesium, Outcomes, and the Effect of Empagliflozin in Heart Failure With Mildly Reduced and Preserved Ejection Fraction: Findings From EMPEROR-Preserved. JACC Heart Fail. 2026 Feb;14(2):102889. doi: 10.1016/j.jchf.2025.102889. Epub 2026 Jan 5. PMID 41493412
- [Derived] Carson P, Teerlink JR, Komajda M, Anand I, Packer M, Butler J, Doehner W, Ferreira JP, Filippatos G, Haass M, Miller A, Pehrson S, Pocock SJ, Iwata T, Brueckmann M, Gasior T, Zannad F, Anker SD. Comparison of Investigator-Reported and Centrally Adjudicated Heart Failure Outcomes in the EMPEROR-Preserved Trial. JACC Heart Fail. 2025 May;13(5):710-721. doi: 10.1016/j.jchf.2024.10.021. Epub 2025 Jan 29. PMID 39895437
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Ferreira JP, Packer M, Sattar N, Butler J, Pocock SJ, Anker SD, Maldonado SG, Panova-Noeva M, Sumin M, Masson S, Zannad F, Januzzi JL. Carbohydrate antigen 125 concentrations across the ejection fraction spectrum in chronic heart failure: The EMPEROR programme. Eur J Heart Fail. 2024 Apr;26(4):788-802. doi: 10.1002/ejhf.3166. Epub 2024 Mar 4. PMID 38439582
- [Derived] Zannad F, Macari S. Drug treatment with empagliflozin was beneficial in people with heart failure with preserved ejection fraction: plain language summary of the EMPEROR-Preserved study. Future Cardiol. 2023 Nov;19(14):671-677. doi: 10.2217/fca-2023-0091. Epub 2023 Nov 9. PMID 37942723
- [Derived] Packer M, Butler J, Zeller C, Pocock SJ, Brueckmann M, Ferreira JP, Filippatos G, Usman MS, Zannad F, Anker SD. Blinded Withdrawal of Long-Term Randomized Treatment With Empagliflozin or Placebo in Patients With Heart Failure. Circulation. 2023 Sep 26;148(13):1011-1022. doi: 10.1161/CIRCULATIONAHA.123.065748. Epub 2023 Aug 24. PMID 37621153
- [Derived] Butler J, Usman MS, Filippatos G, Ferreira JP, Bohm M, Brueckmann M, Januzzi JL, Kaul S, Pina IL, Ponikowski P, Senni M, Sumin M, Verma S, Zaremba-Pechmann L, Pocock SJ, Packer M, Anker S. Safety and Efficacy of Empagliflozin and Diuretic Use in Patients with Heart Failure and Preserved Ejection Fraction: A Post Hoc Analysis of the EMPEROR-Preserved Trial. JAMA Cardiol. 2023 Jul 1;8(7):640-649. doi: 10.1001/jamacardio.2023.1090. PMID 37223933
- [Derived] Bhm M, Anker S, Mahfoud F, Lauder L, Filippatos G, Ferreira JP, Pocock SJ, Brueckmann M, Saloustros I, Schler E, Wanner C, Zannad F, Packer M, Butler J. Empagliflozin, irrespective of blood pressure, improves outcomes in heart failure with preserved ejection fraction: the EMPEROR-Preserved trial. Eur Heart J. 2023 Feb 1;44(5):396-407. doi: 10.1093/eurheartj/ehac693. PMID 36478225
- [Derived] Ferreira JP, Zannad F, Butler J, Filippatos G, Pocock SJ, Brueckmann M, Steubl D, Schueler E, Anker SD, Packer M. Association of Empagliflozin Treatment With Albuminuria Levels in Patients With Heart Failure: A Secondary Analysis of EMPEROR-Pooled. JAMA Cardiol. 2022 Nov 1;7(11):1148-1159. doi: 10.1001/jamacardio.2022.2924. PMID 36129693
- [Derived] Butler J, Filippatos G, Siddiqi TJ, Ferreira JP, Brueckmann M, Bocchi E, Bohm M, Chopra VK, Giannetti N, Iwata T, Januzzi JL, Kaul S, Pina IL, Ponikowski P, Rauch-Krohnert U, Shah SJ, Senni M, Sumin M, Verma S, Zhang J, Pocock SJ, Zannad F, Packer M, Anker SD. Effects of Empagliflozin in Women and Men With Heart Failure and Preserved Ejection Fraction. Circulation. 2022 Oct 4;146(14):1046-1055. doi: 10.1161/CIRCULATIONAHA.122.059755. Epub 2022 Sep 13. PMID 36098051
- [Derived] Zannad F, Ferreira JP, Butler J, Filippatos G, Januzzi JL, Sumin M, Zwick M, Saadati M, Pocock SJ, Sattar N, Anker SD, Packer M. Effect of empagliflozin on circulating proteomics in heart failure: mechanistic insights into the EMPEROR programme. Eur Heart J. 2022 Dec 21;43(48):4991-5002. doi: 10.1093/eurheartj/ehac495. PMID 36017745
- [Derived] Filippatos G, Butler J, Farmakis D, Zannad F, Ofstad AP, Ferreira JP, Green JB, Rosenstock J, Schnaidt S, Brueckmann M, Pocock SJ, Packer M, Anker SD; EMPEROR-Preserved Trial Committees and Investigators. Empagliflozin for Heart Failure With Preserved Left Ventricular Ejection Fraction With and Without Diabetes. Circulation. 2022 Aug 30;146(9):676-686. doi: 10.1161/CIRCULATIONAHA.122.059785. Epub 2022 Jun 28. PMID 35762322
- [Derived] Ferreira JP, Zannad F, Butler J, Filipattos G, Ritter I, Schuler E, Kraus BJ, Pocock SJ, Anker SD, Packer M. Empagliflozin and serum potassium in heart failure: an analysis from EMPEROR-Pooled. Eur Heart J. 2022 Aug 14;43(31):2984-2993. doi: 10.1093/eurheartj/ehac306. PMID 35687107
- [Derived] Januzzi JL Jr, Butler J, Zannad F, Filippatos G, Ferreira JP, Pocock SJ, Sattar N, Verma S, Vedin O, Iwata T, Brueckmann M, Packer M, Anker SD; EMPEROR-Preserved Trial Study Group. Prognostic Implications of N-Terminal Pro-B-Type Natriuretic Peptide and High-Sensitivity Cardiac Troponin T in EMPEROR-Preserved. JACC Heart Fail. 2022 Jul;10(7):512-524. doi: 10.1016/j.jchf.2022.05.004. Epub 2022 Jun 1. PMID 35670067
- [Derived] Vaduganathan M, Claggett BL, Inciardi RM, Fonarow GC, McMurray JJV, Solomon SD. Estimating the Benefits of Combination Medical Therapy in Heart Failure With Mildly Reduced and Preserved Ejection Fraction. Circulation. 2022 Jun 7;145(23):1741-1743. doi: 10.1161/CIRCULATIONAHA.121.058929. Epub 2022 May 23. No abstract available. PMID 35603667
- [Derived] Ferreira JP, Butler J, Zannad F, Filippatos G, Schueler E, Steubl D, Zeller C, Januzzi JL, Pocock S, Packer M, Anker SD. Mineralocorticoid Receptor Antagonists and Empagliflozin in Patients With Heart Failure and Preserved Ejection Fraction. J Am Coll Cardiol. 2022 Mar 29;79(12):1129-1137. doi: 10.1016/j.jacc.2022.01.029. PMID 35331406
- [Derived] Butler J, Filippatos G, Jamal Siddiqi T, Brueckmann M, Bohm M, Chopra VK, Pedro Ferreira J, Januzzi JL, Kaul S, Pina IL, Ponikowski P, Shah SJ, Senni M, Vedin O, Verma S, Peil B, Pocock SJ, Zannad F, Packer M, Anker SD. Empagliflozin, Health Status, and Quality of Life in Patients With Heart Failure and Preserved Ejection Fraction: The EMPEROR-Preserved Trial. Circulation. 2022 Jan 18;145(3):184-193. doi: 10.1161/CIRCULATIONAHA.121.057812. Epub 2021 Nov 15. PMID 34779658
- [Derived] Kanie T, Mizuno A, Takaoka Y, Suzuki T, Yoneoka D, Nishikawa Y, Tam WWS, Morze J, Rynkiewicz A, Xin Y, Wu O, Providencia R, Kwong JS. Dipeptidyl peptidase-4 inhibitors, glucagon-like peptide 1 receptor agonists and sodium-glucose co-transporter-2 inhibitors for people with cardiovascular disease: a network meta-analysis. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD013650. doi: 10.1002/14651858.CD013650.pub2. PMID 34693515
- [Derived] Anker SD, Butler J, Filippatos G, Ferreira JP, Bocchi E, Bohm M, Brunner-La Rocca HP, Choi DJ, Chopra V, Chuquiure-Valenzuela E, Giannetti N, Gomez-Mesa JE, Janssens S, Januzzi JL, Gonzalez-Juanatey JR, Merkely B, Nicholls SJ, Perrone SV, Pina IL, Ponikowski P, Senni M, Sim D, Spinar J, Squire I, Taddei S, Tsutsui H, Verma S, Vinereanu D, Zhang J, Carson P, Lam CSP, Marx N, Zeller C, Sattar N, Jamal W, Schnaidt S, Schnee JM, Brueckmann M, Pocock SJ, Zannad F, Packer M; EMPEROR-Preserved Trial Investigators. Empagliflozin in Heart Failure with a Preserved Ejection Fraction. N Engl J Med. 2021 Oct 14;385(16):1451-1461. doi: 10.1056/NEJMoa2107038. Epub 2021 Aug 27. PMID 34449189
- [Derived] Nassif ME, Kosiborod M. Effects of sodium glucose cotransporter type 2 inhibitors on heart failure. Diabetes Obes Metab. 2019 Apr;21 Suppl 2:19-23. doi: 10.1111/dom.13678. PMID 31081589
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomised, double-blind trial to demonstrate superiority of empagliflozin versus placebo in patients with symptomatic, chronic heart failure and preserved left ventricular ejection fraction (LVEF>40%) under stable treatment of heart failure symptoms.
Pre-assignment Details: Patients were included in the trial after they had signed the informed consent form (ICF). Patients who met all of the inclusion and none of the exclusion criteria were to be included in the trial. All patients were informed that they were free to withdraw their consent at any time during the trial without penalty or prejudice.
Groups:
- Placebo: 1 film-coated tablet of matching placebo was administered orally once daily in patients with chronic heart failure with preserved ejection fraction (HFpEF).
- 10 mg Empagliflozin: 1 film-coated tablet of 10 milligram (mg) of empagliflozin was administered orally once daily in patients with chronic heart failure with preserved ejection fraction (HFpEF).
Period: Overall Study
Arm/Group | Placebo | 10 mg Empagliflozin
Started (Randomised) | 2991 | 2997
Treated | 2989 | 2996
Completed (Patients who did not prematurely discontinue from trial medication) | 2046 | 2051
Not Completed | 945 | 946
Not completed — Adverse Event | 553 | 575
Not completed — Protocol Violation | 30 | 24
Not completed — Lost to Follow-up | 6 | 16
Not completed — Patient refusal to continue, not due to AE | 304 | 284
Not completed — Study drug stopped, reason missing | 6 | 1
Not completed — Medical advice | 6 | 2
Not completed — Due to Covid-19 Pandemic | 2 | 8
Not completed — Investigator decision | 2 | 0
Not completed — Patient decision | 5 | 2
Not completed — Not attending study visits | 3 | 0
Not completed — Patient moved away | 3 | 4
Not completed — Other reason than stated above | 23 | 29
Not completed — Not treated | 2 | 1

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS), including all randomised patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg Empagliflozin | Total
Number analyzed (Participants) | 2991 | 2997 | 5988
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.9 (9.6) | 71.8 (9.3) | 71.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1338 | 1338 | 2676
  Male | 1653 | 1659 | 3312
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 754 | 770 | 1524
  Not Hispanic or Latino | 2236 | 2227 | 4463
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 104 | 90 | 194
  Asian | 411 | 413 | 824
  Native Hawaiian or Other Pacific Islander | 19 | 14 | 33
  Black or African American | 125 | 133 | 258
  White | 2256 | 2286 | 4542
  More than one race | 75 | 60 | 135
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to First Event of Adjudicated Cardiovascular (CV) Death or Adjudicated Hospitalisation for Heart Failure (HHF)
Description: Failure with preserved Ejection Fraction (HFpEF). The incidence rate per 100 patient years (pt-yrs) is presented and calculated as followed:
  Incidence rate per 100 pt-yrs = 100 * number of patients with event / time at risk [years].
  Time at risk [years] = Sum of time at risk [days] over all patients in a treatment group / 365.25.
  Patients without a specific endpoint event were censored at the last date the patient was known to be free of the event or at the end of the planned treatment period, whichever was earlier.
Time Frame: From randomization until completion of the planned treatment phase, up to 1403 days.
Population: Randomised Set (RS), including all randomised patients.
Measure: Number (95% Confidence Interval); unit: Patients with event/100 pt-yrs at risk
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 2991 | 2997
Patients with event/100 pt-yrs at risk | 8.67 [7.94 to 9.44] | 6.86 [6.22 to 7.54]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Cox regression, with terms for treatment, region, baseline status of diabetes, age, sex, left ventricular ejection fraction (LVEF) and glomerular filtration rate estimated by the chronic kidney disease epidemiology collaboration formula with serum creatinine measurement (eGFR (CKD-EPI)cr) at baseline. alpha=0.0497 (resulting from interim analysis); Test type: Superiority — H0: There is no difference between the effect of placebo and the effect of empagliflozin; p = 0.0003, Regression, Cox; Hazard Ratio (HR) = 0.79, 95.03% CI 2-sided [0.69 to 0.90] — Comparison vs. Placebo [T/P]

2. Secondary Outcome: Occurrence of Adjudicated Hospitalisation for Heart Failure (HHF) (First and Recurrent)
Description: Reported is the total number of adjudicated HHF events (first and recurrent) which occurred.
Time Frame: From randomization until completion of the planned treatment phase, up to 1403 days.
Population: Randomised Set (RS), including all randomised patients.
Measure: Number; unit: HHF events
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 2991 | 2997
HHF events | 541 | 407
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Joint frailty model that accounts for dependence between recurrent HHF and cardiovascular death, with terms for age, baseline eGFR (CKD-EPK)cr, baseline LVEF, region, baseline diabetes status, sex, and treatment. eGFR (CKP-EPI)cr: Glomerular filtration rate estimated by the chronic kidney disease epidemiology collaboration formula with serum creatinine measurement LVEF: Left ventricular ejection fraction. alpha=0.0497 (resulting from interim analysis); Test type: Superiority — H0: There is no difference between the effect of placebo and the effect of empagliflozin; p = 0.0009, Joint frailty model; Hazard Ratio (HR) = 0.73, 95.03% CI 2-sided [0.61 to 0.88] — Comparison vs. Placebo [T/P]

3. Secondary Outcome: eGFR (CKD-EPI) cr Slope of Change From Baseline
Description: Glomerular filtration rate estimated by the chronic kidney disease epidemiology collaboration formula with serum creatinine measurement (eGFR(CKD-EPI)cr) slope of change from baseline.
  Available on-treatment change-from-baseline data were used. The slope represents the long term effect of eGFR change from baseline and provides the yearly rate of decline.
  Timepoints after baseline were included in calculation of slope of change from baseline.
  The slope per patient was calculated using a random coefficient model with terms for treatment, region, baseline status of diabetes, age, sex, left ventricular ejection fraction (LVEF) and glomerular filtration rate estimated by the chronic kidney disease epidemiology collaboration formula (eGFR (CKD-EPI)cr) at baseline and in addition the factors "time", "treatment-by-time interaction", and "baseline eGFR (CKD-EPI)cr-by-time interaction".
Time Frame: At baseline, week 4, 12, 32, 52, 76, 100, 124, 148, 172 and week 196, up to 1043 days.
Population: Only patients included in the treated set (TS) and with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: mL/min/ 1.73 meters squared/year
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 2911 | 2925
mL/min/ 1.73 meters squared/year | -2.616 (0.108) | -1.253 (0.108)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Random coefficient model allowing for random intercept and random slope per patient, with factors age, baseline eGFR (CKD-EPI), baseline LVEF as linear covariate(s) and region, baseline diabetes status, sex, baseline-by-time interaction, treatment-by-time interaction and treatment as fixed effects. Only 'on-treatment' data from treated patients were used. alpha=0.001. covariance structure: Unstructured; Test type: Superiority — H0: There is no difference between the effect of placebo and the effect of empagliflozin; p < 0.0001, Random intercept random coeff. model; Treatment by time interaction = 1.363, 99.9% CI 2-sided [0.861 to 1.865] — Empa 10 mg vs. Placebo slope [/year]

4. Secondary Outcome: Time to the First Event in the Composite Renal Endpoint: Chronic Dialysis, Renal Transplant, or Sustained Reduction in eGFR (CKD-EPI)cr
Description: Chronic dialysis was defined as dialysis with a frequency of twice per week or more for at least 90 days.
  Sustained was determined by two or more consecutive post-baseline central laboratory measurement separated by at least 30 days.
  Reduction in glomerular filtration rate estimated by the chronic kidney disease epidemiology collaboration formula with serum creatinine measurement (eGFR (CKD-EPI)cr) was defined as reduction in eGFR from baseline ≥40%, eGFR <15 mL/min/1.73 m^2 for patients with baseline eGFR ≥30 mL/min/1.73 m^2, or eGFR <10 mL/min/1.73 m^2 for patients with baseline eGFR <30 mL/min/1.73 m^2.
  The incidence rate per 100 patient years (100 * number of patients with event / time at risk [years]) is reported. Time at risk [year] is calculated as: Sum of time at risk [days] over all patients in a treatment group / 365.25.
  Abbreviation:
  Patient-years (pt-yrs).
Time Frame: From randomization until completion of the planned treatment phase, up to 1403 days.
Population: Randomised Set (RS), including all randomised patients.
Measure: Number (95% Confidence Interval); unit: Patients with event /100 pt-yrs at risk
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 2991 | 2997
Patients with event /100 pt-yrs at risk | 2.23 [1.84 to 2.66] | 2.13 [1.74 to 2.54]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Cox regression model included terms age, baseline glomerular filtration rate estimated by the chronic kidney disease epidemiology collaboration formula with serum creatinine measurement (eGFR (CKD-EPI)cr), region, baseline diabetes status, sex, baseline Left ventricular ejection fraction (LVEF) and treatment; Test type: Other; p = 0.7243, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.73 to 1.24] — Comparison vs Placebo [T/P]

5. Secondary Outcome: Time to First Adjudicated Hospitalisation for Heart Failure (HHF)
Description: Time to first adjudicated HHF. The incidence rate per 100 patient years (pt-yrs) is presented and calculated as followed:
  Incidence rate per 100 pt-yrs = 100 * number of patients with event / time at risk [years].
  Time at risk [years] = Sum of time at risk [days] over all patients in a treatment group / 365.25.
  Patients without a specific endpoint event were censored at the last date the patient was known to be free of the event or at the end of the planned treatment period, whichever was earlier.
Time Frame: From randomization until completion of the planned treatment phase, up to 1403 days.
Population: Randomised Set (RS), including all randomised patients.
Measure: Number (95% Confidence Interval); unit: Patients with event /100 pt-yrs at risk
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 2991 | 2997
Patients with event /100 pt-yrs at risk | 5.97 [5.37 to 6.62] | 4.28 [3.78 to 4.82]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; [analysis description as in outcome 4, analysis 1]; Test type: Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.60 to 0.83] — Comparison vs. Placebo [T/P]

6. Secondary Outcome: Time to Adjudicated Cardiovascular (CV) Death
Description: Time to adjudicated CV death. The incidence rate per 100 patient years (pt-yrs) is presented and calculated as followed:
  Incidence rate per 100 pt-yrs = 100 * number of patients with event / time at risk [years].
  Time at risk [years] = Sum of time at risk [days] over all patients in a treatment group / 365.25.
  Patients without a specific endpoint event were censored at the last date the patient was known to be free of the event or at the end of the planned treatment period, whichever was earlier.
Time Frame: From randomization until completion of the planned treatment phase, up to 1403 days.
Population: Randomised Set (RS), including all randomised patients.
Measure: Number (95% Confidence Interval); unit: Patients with event /100 pt-yrs at risk
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 2991 | 2997
Patients with event /100 pt-yrs at risk | 3.81 [3.35 to 4.31] | 3.42 [2.98 to 3.89]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.2951, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.76 to 1.09] — Comparison vs. Placebo [T/P]

7. Secondary Outcome: Time to All-cause Mortality
Description: Time to all-cause mortality. The incidence rate per 100 patient years (pt-yrs) is presented and calculated as followed:
  Incidence rate per 100 pt-yrs = 100 * number of patients with event / time at risk [years].
  Time at risk [years] = Sum of time at risk [days] over all patients in a treatment group / 365.25.
  Patients without a specific endpoint event were censored at the last date the patient was known to be free of the event or at the end of the planned treatment period, whichever was earlier.
Time Frame: From randomization until completion of the planned treatment phase, up to 1403 days.
Population: Randomised Set (RS), including all randomised patients.
Measure: Number (95% Confidence Interval); unit: Patients with event /100 pt-yrs at risk
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 2991 | 2997
Patients with event /100 pt-yrs at risk | 6.67 [6.05 to 7.32] | 6.60 [5.98 to 7.24]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.9893, Regression, Cox; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.87 to 1.15] — Comparison vs. Placebo [T/P]

8. Secondary Outcome: Time to Onset of Diabetes Mellitus (DM) in Patients With Pre-DM
Description: Time to onset of DM (defined as HbA1c ≥6.5% or as diagnosed by the investigator) in patients with pre-DM.
  Pre-DM was defined as no history of DM and no HbA1c ≥6.5% before treatment, and a pre-treatment HbA1c value of ≥5.7% and <6.5%.
  The incidence rate per 100 patient years (pt-yrs) is presented and calculated as followed:
  Incidence rate per 100 pt-yrs = 100 * number of patients with event / time at risk [years].
  Time at risk [years] = Sum of time at risk [days] over all patients in a treatment group / 365.25.
  Patients without a specific endpoint event were censored at the last date the patient was known to be free of the event or at the end of the planned treatment period, whichever was earlier.
Time Frame: From randomization until completion of the planned treatment phase, to 1403 days.
Population: Randomised Set (RS), including all randomised patients and with available data for this endpoint.
Measure: Number (95% Confidence Interval); unit: Patients with event /100 pt-yrs at risk
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 979 | 1001
Patients with event /100 pt-yrs at risk | 7.39 [6.21 to 8.68] | 6.12 [5.07 to 7.26]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.1539, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.65 to 1.07] — Comparison vs. Placebo [T/P]

9. Secondary Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionaire (KCCQ) Clinical Summary Score at Week 52
Description: The KCCQ is a 23-item self-administered questionnaire designed to evaluate physical limitations, symptoms (frequency, severity, and changes over time), social limitations, self-efficacy, and quality of life in patients with Heart Failure. The KCCQ-clinical summary score comprises the following domains: Symptom frequency, symptom burden and physical limitation. The score is calculated by summing domain responses and then transforming scores to a 0-100 unit scale with higher scores indicating better health status.
  For patients who died, a worst score (score of 0) was imputed for the score at all subsequent scheduled visits after the date of death where the score would have been assessed.
  Change from baseline in KCCQ-score at week 52 was modeled using a MMRM with visit (week 12, 32 and 52) as repeated measures, adjusted mean (standard error) at week 52 is reported.
Time Frame: At baseline and at week 12, week 32 and week 52.
Population: Only Patients included in the treated set (TS) including values obtained on treatment. The number of patients analysed displays the number of patients with available data at the timepoint of interests.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 2335 | 2333
Score on a scale | 3.18 (0.31) | 4.51 (0.31)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Model includes age, baseline glomerular filtration rate estimated by the chronic kidney disease epidemiology collaboration formula (eGFR (CKD-EPI)), baseline Left ventricular ejection fraction (LVEF) as linear covariate(s) and region, baseline diabetes status, sex, week reachable, treatment-by-visit interaction, baseline KCCQ-Clinical-Summary-Score-by-visit interaction as fixed effect(s). Unstructured covariance structure; Test type: Other; p = 0.0028, Mixed Model Repeated Measures (MMRM); Adjusted mean difference = 1.32, 95% CI 2-sided [0.45 to 2.19], Standard Error of Mean 0.44 — Comparison vs Placebo [T-P]

10. Secondary Outcome: Occurrence of All-cause Hospitalisation (First and Recurrent)
Description: Occurrence of all-cause hospitalisation (first and recurrent). Total number of all cause hospitalisations is reported.
Time Frame: From randomization until completion of the planned treatment phase, up to 1403 days.
Population: Randomised Set (RS), including all randomised patients.
Measure: Number; unit: Events of all-cause hospitialisations
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 2991 | 2997
Events of all-cause hospitialisations | 2769 | 2566
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Joint frailty model that accounts for the dependence between recurrent all-cause hospitalisation and all-cause mortality was used. Joint frailty model with terms for age, baseline glomerular filtration rate estimated by the chronic kidney disease epidemiology collaboration formula (eGFR (CKD-EPI)), baseline Left ventricular ejection fraction (LVEF), treatment, region, baseline diabetes status and sex; Test type: Other; p = 0.1012, Joint frailty model; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.85 to 1.01] — Comparison vs. Placebo [T/P]

ADVERSE EVENTS:
Time Frame: [All-cause Mortality]: From study start until end of study, up to 1438 days. [Serious adverse events (AE) and other AE]:From time of the first drug intake until 7 days (Residual Effect Period) after the last drug intake, up to 1410 days.
Description: [All-cause mortality]: Randomised Set (RS), including all randomised patients. [Serious AE and other AE]: Treated Set (TS), including all patients treated with at least one dose of the study medication.
Arm/Group | Placebo | 10 mg Empagliflozin
All-Cause Mortality (participants affected / at risk) | 427/2991 | 422/2997
Serious Adverse Events (participants affected / at risk) | 1543/2989 | 1436/2996
Other Adverse Events (participants affected / at risk) | 1274/2989 | 1191/2996
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2989) | 10 mg Empagliflozin (N=2996)
Anaemia (Blood and lymphatic system disorders) | 30 | 19
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 4 | 2
Coagulopathy (Blood and lymphatic system disorders) | 2 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 12 | 6
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 4 | 2
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 8
Acute left ventricular failure (Cardiac disorders) | 4 | 4
Acute myocardial infarction (Cardiac disorders) | 48 | 50
Adams-Stokes syndrome (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 23 | 28
Angina unstable (Cardiac disorders) | 23 | 26
Aortic valve incompetence (Cardiac disorders) | 1 | 4
Aortic valve stenosis (Cardiac disorders) | 4 | 4
Arrhythmia (Cardiac disorders) | 5 | 2
Arrhythmia supraventricular (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 80 | 92
Atrial flutter (Cardiac disorders) | 21 | 14
Atrial tachycardia (Cardiac disorders) | 3 | 2
Atrial thrombosis (Cardiac disorders) | 2 | 1
Atrioventricular block (Cardiac disorders) | 2 | 2
Atrioventricular block complete (Cardiac disorders) | 5 | 11
Atrioventricular block second degree (Cardiac disorders) | 2 | 6
Bradyarrhythmia (Cardiac disorders) | 1 | 2
Bradycardia (Cardiac disorders) | 6 | 6
Bundle branch block left (Cardiac disorders) | 1 | 0
Bundle branch block right (Cardiac disorders) | 1 | 1
Cardiac amyloidosis (Cardiac disorders) | 3 | 2
Cardiac arrest (Cardiac disorders) | 8 | 12
Cardiac failure (Cardiac disorders) | 594 | 448
Cardiac failure acute (Cardiac disorders) | 29 | 12
Cardiac failure chronic (Cardiac disorders) | 30 | 25
Cardiac failure congestive (Cardiac disorders) | 66 | 57
Cardiac sarcoidosis (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 2 | 5
Cardiogenic shock (Cardiac disorders) | 12 | 5
Cardiopulmonary failure (Cardiac disorders) | 2 | 2
Cardiorenal syndrome (Cardiac disorders) | 1 | 2
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Chronic left ventricular failure (Cardiac disorders) | 0 | 2
Chronotropic incompetence (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 32 | 22
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 3 | 3
Coronary artery stenosis (Cardiac disorders) | 8 | 4
Ischaemic cardiomyopathy (Cardiac disorders) | 3 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 7 | 4
Mitral valve stenosis (Cardiac disorders) | 0 | 3
Myocardial infarction (Cardiac disorders) | 27 | 37
Myocardial ischaemia (Cardiac disorders) | 9 | 8
Myocardial necrosis (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 1
Prinzmetal angina (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 3 | 1
Silent myocardial infarction (Cardiac disorders) | 0 | 1
Sinoatrial block (Cardiac disorders) | 1 | 1
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 7
Sinus node dysfunction (Cardiac disorders) | 8 | 8
Stress cardiomyopathy (Cardiac disorders) | 3 | 0
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 3 | 3
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Torsade de pointes (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 3 | 2
Ventricular arrhythmia (Cardiac disorders) | 1 | 1
Ventricular dyskinesia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 3 | 0
Ventricular failure (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 4 | 5
Ventricular tachycardia (Cardiac disorders) | 22 | 22
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Buried penis syndrome (Congenital, familial and genetic disorders) | 1 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 2
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 3 | 0
Phimosis (Congenital, familial and genetic disorders) | 3 | 4
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 1
Talipes (Congenital, familial and genetic disorders) | 0 | 1
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 2 | 0
Deafness bilateral (Ear and labyrinth disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 2 | 5
Deafness unilateral (Ear and labyrinth disorders) | 4 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Mixed deafness (Ear and labyrinth disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 2 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 4 | 2
Vertigo positional (Ear and labyrinth disorders) | 0 | 4
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Basedow's disease (Endocrine disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 3
Hyperplasia adrenal (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 2
Pituitary apoplexy (Endocrine disorders) | 0 | 1
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 | 0
Amaurosis fugax (Eye disorders) | 2 | 1
Blindness transient (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 10 | 10
Cataract nuclear (Eye disorders) | 2 | 1
Conjunctival disorder (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 10 | 8
Macular degeneration (Eye disorders) | 2 | 3
Macular fibrosis (Eye disorders) | 1 | 2
Macular hole (Eye disorders) | 1 | 1
Macular ischaemia (Eye disorders) | 0 | 1
Neovascular age-related macular degeneration (Eye disorders) | 1 | 0
Normal tension glaucoma (Eye disorders) | 1 | 1
Open angle glaucoma (Eye disorders) | 3 | 2
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Retinal artery embolism (Eye disorders) | 2 | 0
Retinal artery occlusion (Eye disorders) | 1 | 2
Retinal detachment (Eye disorders) | 2 | 1
Retinal ischaemia (Eye disorders) | 1 | 0
Retinal tear (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 4 | 2
Visual acuity reduced (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 2
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 2 | 4
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 4
Diverticular perforation (Gastrointestinal disorders) | 1 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 | 3
Duodenitis (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Faecal vomiting (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 6 | 4
Gastritis erosive (Gastrointestinal disorders) | 3 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 17 | 14
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal polyp (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhagic ascites (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 4 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 2
Hiatus hernia (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 4 | 3
Ileus paralytic (Gastrointestinal disorders) | 1 | 4
Incarcerated inguinal hernia (Gastrointestinal disorders) | 2 | 2
Incarcerated umbilical hernia (Gastrointestinal disorders) | 2 | 3
Inguinal hernia (Gastrointestinal disorders) | 9 | 8
Intestinal angina (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 3 | 4
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal strangulation (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 4 | 4
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 1
Mechanical ileus (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 1 | 1
Mesenteric artery embolism (Gastrointestinal disorders) | 1 | 0
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 2 | 1
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal rupture (Gastrointestinal disorders) | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatic disorder (Gastrointestinal disorders) | 1 | 0
Pancreatic failure (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 1
Pancreatitis acute (Gastrointestinal disorders) | 2 | 3
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 1
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 5
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Stomach mass (Gastrointestinal disorders) | 0 | 1
Subacute pancreatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 5
Volvulus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 2
Accidental death (General disorders) | 0 | 1
Asthenia (General disorders) | 4 | 1
Cardiac death (General disorders) | 3 | 4
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 6 | 3
Death (General disorders) | 38 | 56
Discomfort (General disorders) | 0 | 1
Drowning (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Fibrosis (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 2
Hernia (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 2 | 0
Inflammation (General disorders) | 0 | 1
Injection site phlebitis (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Medical device site oedema (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 3 | 6
Necrosis (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 16 | 14
Oedema peripheral (General disorders) | 2 | 0
Pacemaker generated arrhythmia (General disorders) | 0 | 1
Physical deconditioning (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 2
Stent-graft endoleak (General disorders) | 1 | 1
Strangulated hernia (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 9 | 4
Sudden death (General disorders) | 8 | 10
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Vascular stent occlusion (General disorders) | 1 | 0
Vascular stent stenosis (General disorders) | 1 | 1
Vessel puncture site bruise (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 4 | 6
Biliary colic (Hepatobiliary disorders) | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 2
Cardiac cirrhosis (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 3
Cholangitis acute (Hepatobiliary disorders) | 1 | 3
Cholecystitis (Hepatobiliary disorders) | 6 | 6
Cholecystitis acute (Hepatobiliary disorders) | 3 | 4
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 7 | 6
Cholestasis (Hepatobiliary disorders) | 2 | 1
Cholestatic liver injury (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 6 | 7
Hepatic failure (Hepatobiliary disorders) | 2 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 3
Hepatitis acute (Hepatobiliary disorders) | 0 | 3
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0
Hepatorenal failure (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 2 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Liver disorder (Hepatobiliary disorders) | 3 | 2
Liver injury (Hepatobiliary disorders) | 9 | 7
Allergy to vaccine (Immune system disorders) | 1 | 0
Amyloidosis (Immune system disorders) | 0 | 2
Anaphylactic reaction (Immune system disorders) | 1 | 0
Corneal graft rejection (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Abdominal sepsis (Infections and infestations) | 1 | 3
Abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 2 | 1
Abscess neck (Infections and infestations) | 1 | 0
Acinetobacter infection (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 5 | 4
Arthritis bacterial (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 2 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial food poisoning (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 3 | 1
Bacterial translocation (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 1 | 0
Breast cellulitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 12 | 4
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bullous erysipelas (Infections and infestations) | 0 | 1
Bursitis infective (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 47 | 49
COVID-19 pneumonia (Infections and infestations) | 17 | 25
Cardiac valve abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 8 | 22
Cholangitis infective (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Clostridial sepsis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 5 | 0
Clostridium difficile infection (Infections and infestations) | 3 | 1
Colon gangrene (Infections and infestations) | 1 | 0
Complicated appendicitis (Infections and infestations) | 1 | 0
Coronavirus infection (Infections and infestations) | 3 | 2
Cystitis (Infections and infestations) | 2 | 2
Dengue fever (Infections and infestations) | 1 | 3
Device related infection (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 2 | 0
Diabetic gangrene (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 5 | 6
Dysentery (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 3 | 5
Endocarditis bacterial (Infections and infestations) | 0 | 2
Endocarditis staphylococcal (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1
Enterobacter sepsis (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 4 | 5
Escherichia sepsis (Infections and infestations) | 1 | 0
Fournier's gangrene (Infections and infestations) | 0 | 1
Fungal oesophagitis (Infections and infestations) | 1 | 0
Gallbladder empyema (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 4 | 4
Gastroenteritis (Infections and infestations) | 7 | 8
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 1 | 0
Hepatitis A (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 3
Herpes zoster infection neurological (Infections and infestations) | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1
Infected gouty tophus (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 2
Infectious pleural effusion (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 5 | 2
Intervertebral discitis (Infections and infestations) | 4 | 0
Intestinal sepsis (Infections and infestations) | 0 | 2
Joint abscess (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Large intestine infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 2 | 2
Localised infection (Infections and infestations) | 2 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Ludwig angina (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 2 | 1
Meningitis bacterial (Infections and infestations) | 1 | 0
Neurocysticercosis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 5 | 6
Osteomyelitis acute (Infections and infestations) | 0 | 1
Parotid abscess (Infections and infestations) | 1 | 0
Pathogen resistance (Infections and infestations) | 0 | 1
Perineal abscess (Infections and infestations) | 1 | 1
Periodontitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 3 | 2
Peritonitis bacterial (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 1
Peritonsillitis (Infections and infestations) | 1 | 0
Petrositis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 119 | 100
Pneumonia bacterial (Infections and infestations) | 8 | 6
Pneumonia parainfluenzae viral (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 3 | 0
Postoperative abscess (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 2 | 3
Prostatitis Escherichia coli (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 4 | 5
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 3
Pyelonephritis acute (Infections and infestations) | 3 | 7
Respiratory tract infection (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 21 | 26
Septic shock (Infections and infestations) | 11 | 11
Severe acute respiratory syndrome (Infections and infestations) | 2 | 0
Severe fever with thrombocytopenia syndrome (Infections and infestations) | 1 | 0
Small intestine gangrene (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 2 | 1
Staphylococcal sepsis (Infections and infestations) | 3 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Superinfection (Infections and infestations) | 1 | 0
Suspected COVID-19 (Infections and infestations) | 2 | 0
Systemic bacterial infection (Infections and infestations) | 0 | 2
Systemic candida (Infections and infestations) | 1 | 0
Testicular abscess (Infections and infestations) | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 28 | 36
Urosepsis (Infections and infestations) | 12 | 12
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0
Wound abscess (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 3 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Wound sepsis (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 4
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Bursa injury (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 3 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Corneal graft failure (Injury, poisoning and procedural complications) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 4
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Deafness traumatic (Injury, poisoning and procedural complications) | 0 | 1
Diffuse axonal injury (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 1
Dural tear (Injury, poisoning and procedural complications) | 0 | 1
Epidural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 30 | 31
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 1
Femur fracture (Injury, poisoning and procedural complications) | 12 | 14
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 2 | 1
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 1
Genital contusion (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 4 | 3
Heart injury (Injury, poisoning and procedural complications) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 7 | 9
Humerus fracture (Injury, poisoning and procedural complications) | 5 | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 2
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 4 | 1
Maisonneuve fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 7 | 3
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Post procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 | 0
Postoperative delirium (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Procedural shock (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 2
Radius fracture (Injury, poisoning and procedural complications) | 1 | 2
Rib fracture (Injury, poisoning and procedural complications) | 3 | 6
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 3
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 2 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 3
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 2
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 4 | 8
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 4 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 3
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 2 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1
Traumatic spinal cord compression (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Urethral injury (Injury, poisoning and procedural complications) | 2 | 0
Urethral stricture postoperative (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 6 | 4
Anticoagulation drug level below therapeutic (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood ketone body increased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 2
Blood urine present (Investigations) | 1 | 0
Brain natriuretic peptide (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 4 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 3 | 1
Liver function test abnormal (Investigations) | 2 | 0
Occult blood positive (Investigations) | 1 | 0
Prostatic specific antigen abnormal (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 2
Weight decreased (Investigations) | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 8 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 15 | 5
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 | 0
Diabetic complication (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 3
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 18 | 11
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Food intolerance (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 5 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 4
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 20 | 12
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 7 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 3
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 3 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 3 | 1
Ketosis (Metabolism and nutrition disorders) | 2 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 3 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 11 | 6
Obesity (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 | 2
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 3
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 16 | 11
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 9 | 3
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 5 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Sacroiliac joint dysfunction (Musculoskeletal and connective tissue disorders) | 0 | 1
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 3 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral column mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal gland cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 | 17
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glomangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Keratinising squamous cell carcinoma of nasopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 10
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Myxoid liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasopharyngeal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasopharyngeal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Neuroendocrine tumour of the lung metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 11
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Skin cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 7
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the parotid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Altered state of consciousness (Nervous system disorders) | 1 | 2
Arachnoid cyst (Nervous system disorders) | 1 | 0
Brain compression (Nervous system disorders) | 0 | 1
Brain injury (Nervous system disorders) | 3 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Brain stem ischaemia (Nervous system disorders) | 0 | 1
Brain stem stroke (Nervous system disorders) | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 1 | 1
Carotid artery aneurysm (Nervous system disorders) | 0 | 2
Carotid artery disease (Nervous system disorders) | 1 | 0
Carotid artery dissection (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 4 | 3
Carotid artery stenosis (Nervous system disorders) | 4 | 2
Carpal tunnel syndrome (Nervous system disorders) | 0 | 2
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebellar haematoma (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 1 | 1
Cerebral artery occlusion (Nervous system disorders) | 1 | 1
Cerebral atrophy (Nervous system disorders) | 2 | 0
Cerebral disorder (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 3
Cerebral infarction (Nervous system disorders) | 10 | 14
Cerebral ischaemia (Nervous system disorders) | 0 | 2
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 20 | 21
Cervical cord compression (Nervous system disorders) | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 2
Coma (Nervous system disorders) | 0 | 1
Cranial nerve palsies multiple (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 10 | 14
Dementia Alzheimer's type (Nervous system disorders) | 1 | 1
Demyelination (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 6 | 3
Drop attacks (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 4
Encephalomalacia (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 2
Epilepsy (Nervous system disorders) | 3 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 1
Haemorrhagic stroke (Nervous system disorders) | 7 | 7
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 2 | 2
Hemiplegia (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 2
Hydrocephalus (Nervous system disorders) | 0 | 2
Hypertensive encephalopathy (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypoglycaemic seizure (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 3 | 3
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 35 | 42
Lacunar infarction (Nervous system disorders) | 3 | 2
Lacunar stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 1
Lumbar radiculopathy (Nervous system disorders) | 2 | 0
Migraine (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 2 | 0
Neurological symptom (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 3 | 0
Parkinsonism (Nervous system disorders) | 0 | 1
Posterior cortical atrophy (Nervous system disorders) | 0 | 1
Postresuscitation encephalopathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 3
Sciatica (Nervous system disorders) | 2 | 5
Seizure (Nervous system disorders) | 7 | 3
Senile dementia (Nervous system disorders) | 0 | 1
Sensorimotor disorder (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 5 | 0
Syncope (Nervous system disorders) | 19 | 23
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Thoracic radiculopathy (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 21 | 20
Tremor (Nervous system disorders) | 1 | 0
Vascular dementia (Nervous system disorders) | 1 | 1
Vascular encephalopathy (Nervous system disorders) | 1 | 2
Vertebral artery stenosis (Nervous system disorders) | 0 | 1
Vertebral artery thrombosis (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Device breakage (Product Issues) | 0 | 1
Device dislocation (Product Issues) | 1 | 1
Device failure (Product Issues) | 0 | 2
Device leakage (Product Issues) | 0 | 1
Device malfunction (Product Issues) | 0 | 1
Thrombosis in device (Product Issues) | 0 | 1
Adjustment disorder (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 3 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 12 | 9
Depression (Psychiatric disorders) | 1 | 1
Disorientation (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Nosophobia (Psychiatric disorders) | 0 | 1
Paranoia (Psychiatric disorders) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 107 | 81
Bladder tamponade (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 25 | 16
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 3
End stage renal disease (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 3 | 4
Hydronephrosis (Renal and urinary disorders) | 0 | 4
Ketonuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 2
Nephropathy (Renal and urinary disorders) | 1 | 2
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Postrenal failure (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 3
Renal colic (Renal and urinary disorders) | 0 | 5
Renal failure (Renal and urinary disorders) | 21 | 9
Renal impairment (Renal and urinary disorders) | 42 | 38
Renal injury (Renal and urinary disorders) | 2 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 2
Urethral caruncle (Renal and urinary disorders) | 1 | 0
Urethral cyst (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 3
Urinary bladder rupture (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 5 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2
Vesical fistula (Renal and urinary disorders) | 1 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 0
Acquired phimosis (Reproductive system and breast disorders) | 0 | 1
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 8
Cervix disorder (Reproductive system and breast disorders) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Prostatitis (Reproductive system and breast disorders) | 2 | 0
Uterine inflammation (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 20 | 8
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 37 | 23
Combined pulmonary fibrosis and emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 13 | 8
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 | 14
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 3 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 5 | 4
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Paraneoplastic dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1
Peau d'orange (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 11 | 6
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Heart valve replacement (Surgical and medical procedures) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0
Angiodysplasia (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 4 | 1
Aortic aneurysm rupture (Vascular disorders) | 2 | 1
Aortic dissection (Vascular disorders) | 4 | 0
Aortic stenosis (Vascular disorders) | 5 | 7
Aortic thrombosis (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Bleeding varicose vein (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 4 | 3
Cyanosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 12 | 6
Dry gangrene (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 0 | 1
Essential hypertension (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 4 | 2
Femoral artery aneurysm (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 3 | 6
Haemorrhage (Vascular disorders) | 1 | 0
Haemorrhagic infarction (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 12 | 8
Hypertensive crisis (Vascular disorders) | 32 | 13
Hypertensive emergency (Vascular disorders) | 4 | 1
Hypertensive urgency (Vascular disorders) | 5 | 3
Hypotension (Vascular disorders) | 19 | 26
Hypovolaemic shock (Vascular disorders) | 6 | 2
Iliac artery dissection (Vascular disorders) | 0 | 1
Iliac artery occlusion (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 1
Malignant hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 3 | 6
Penetrating aortic ulcer (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 16 | 14
Peripheral artery aneurysm (Vascular disorders) | 1 | 1
Peripheral artery occlusion (Vascular disorders) | 6 | 6
Peripheral artery stenosis (Vascular disorders) | 3 | 2
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 5 | 7
Peripheral vascular disorder (Vascular disorders) | 1 | 2
Peripheral venous disease (Vascular disorders) | 0 | 2
Phlebitis (Vascular disorders) | 1 | 0
Phlebitis superficial (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 2 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 2
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 2 | 0
Vasculitis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2989) | 10 mg Empagliflozin (N=2996)
Anaemia (Blood and lymphatic system disorders) | 164 | 119
Atrial fibrillation (Cardiac disorders) | 156 | 137
Urinary tract infection (Infections and infestations) | 160 | 207
Fall (Injury, poisoning and procedural complications) | 193 | 189
Diabetes mellitus (Metabolism and nutrition disorders) | 200 | 139
Hyperkalaemia (Metabolism and nutrition disorders) | 194 | 170
Hyperuricaemia (Metabolism and nutrition disorders) | 208 | 131
Renal impairment (Renal and urinary disorders) | 181 | 177
Hypertension (Vascular disorders) | 248 | 212
Hypotension (Vascular disorders) | 176 | 212

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT03057951/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT03057951/SAP_001.pdf